CLINICAL TRIAL: NCT00642590
Title: Antioxidant Status, Diet and Early Pregnancy
Brief Title: Lifestyle and Fertility Study on Antioxidant Status, Diet and Early Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Dartmouth-Hitchcock Medical Center (Other); Penn State University (Other); Tufts University (Other); Emory University (Other)
Responsible Party: Sponsor
Other Study IDs: R01HD049762 (NIH)
Record Dates: First submitted 2008-03-21; First posted 2008-03-25 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Infertility; Pregnancy; Fertility; Nutrition; Life Style
Keywords: Fertility; Pregnancy; Conception; Infertility; Behavioral; Lifestyle; Nutrition
MeSH Terms: conditions — Infertility; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma, serum, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Healthy couples who are planning their first pregnancy.

SUMMARY:
Researchers believe that certain lifestyle factors can influence a couple's ability to conceive and have a baby. The ISIS Study will look at the health habits of couples who are planning their first pregnancy, and then attempt to measure the effect these habits have on the couple's fertility. The ISIS Study hopes to clarify the link between lifestyle and fertility, and believes that information gained in this project may help future couples in their attempts to conceive.

DETAILED DESCRIPTION:
Only one-fourth to one-third of fertilized human eggs are likely to survive to produce a term baby. The causes of these reproductive failures are substantially unknown, but scientific evidence suggests that they may, in part, be due to exposures such as pre-conception nutrition, that may result in insults to the oocyte and periconceptual embryo. Early reproductive events may have long-lasting impact as several have recently been identified as antecedents to adult-onset diseases. The goal of this prospective epidemiologic study is to evaluate the hypothesis that increased oxidative stress results in delayed time-to-pregnancy or early pregnancy loss. Recently, reactive oxygen species (ROS) have been associated with spontaneous abortion, preeclampsia, and premature preterm rupture of the membranes in women and defective sperm function in men. In living cells ROS are formed continuously as a consequence of both biochemical reactions and external factors. In this prospective cohort study of healthy couples who are planning pregnancy, we are evaluating time-to-pregnancy, defined as the number of menstrual cycles from the cessation of contraception to a clinically recognized pregnancy, and early unrecognized pregnancy loss. Unrecognized pregnancy and subsequent early loss will be determined by measuring urinary human chorionic gonadotropin (hCG). Diet will be assessed in both partners prior to conception using the Block food frequency questionnaire and serum assays for the antioxidants vitamins C and E, the carotenoids, and selenium. Two urinary biomarkers of oxidative stress, 8-hydroxy-2'-deoxyguanosine and F2a-isoprostanes, and a serum biomarker of antioxidative capacity, oxygen radical absorbance capacity, will be measured in the women. The proposed study has a number of strengths: 1) it is large and prospective in design, with diet and oxidative stress measured prior to conception; 2) a highly sensitive and specific assay for hCG will be used to detect conceptions as early as the time of implantation; 3) dietary intake and biomarker assays of antioxidant status will be assessed twice during the preconception period using state-of-the-art assessment methods including a diet calibration substudy; 4) the proposed research has the potential to fill gaps in our understanding of the role of diet in achieving successful conception, an area where very little investigation has been done.

ELIGIBILITY:
Inclusion Criteria:

* Female is between 18 and 39 years of age
* Female is having regular periods
* Couple is currently using some form of contraception (e.g., oral contraceptives, barrier methods, timing method), but planning to get pregnant in the near future.

Exclusion Criteria:

* Female has a previous pregnancy
* Female has tried for 12 months or more to achieve a pregnancy without success, or has undergone fertility treatment
* Female has received a diagnosis of polycystic ovary syndrome (PCOS)
* Female has another serious medical condition (e.g. heart disease, kidney disease, diabetes, thyroid disease, clinical depression, or an acute chronic infection)
* Male has tried for 12 months or more to achieve a conception without success
* Male has had a fertility related condition (e.g., zoo- or oligospermia, other abnormal semen analysis, cryptorchidism, or testicular cancer)
* Male has another serious medical condition (e.g. heart disease, kidney disease, diabetes, thyroid disease, clinical depression, or an acute chronic infection)

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We are looking for couples who are planning a pregnancy. This must be a first pregnancy for women, ages 18 to 39, and both partners must be in good general health with no history of infertility.
Sampling Method: Non-Probability Sample
Enrollment: 266 (Actual)
Dates: Start 2008-03; Primary Completion 2016-12 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Time to pregnancy | Couples will be followed from preconception to the outcome of pregnancy.
  Time to pregnancy is defined as the number of menstrual cycles from the cessation of contraception to a clinically recognized pregnancy.
Early pregnancy loss | First trimester of pregnancy
  Pregnancy and subsequent early loss will be determined by measuring urinary human chorionic gonadotropin (hCG).

CONTACTS AND LOCATIONS:
Overall Officials: Marlene B. Goldman, MS, ScD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (2):
- United States (2):
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Penn State University, University Park, Pennsylvania

REFERENCES:
- [Background] Ruder EH, Hartman TJ, Blumberg J, Goldman MB. Oxidative stress and antioxidants: exposure and impact on female fertility. Hum Reprod Update. 2008 Jul-Aug;14(4):345-57. doi: 10.1093/humupd/dmn011. Epub 2008 Jun 4. PMID 18535004
- [Background] Paine MA, Ruder EH, Hartman TJ, Blumberg J, Goldman MB. Oxidative stress, oogenesis, and folliculogenesis. In: Studies on Women's Health. Oxidative Stress in Applied Basic Research and Clinical Practice. Agarwal A, Aziz N, Rizk B (eds.), Humana Press, 2013.
- [Background] Ruder EH, Hartman TJ, Goldman MB. Impact of oxidative stress on female fertility. Curr Opin Obstet Gynecol. 2009 Jun;21(3):219-22. doi: 10.1097/gco.0b013e32832924ba. PMID 19469044
- [Background] Darche RL, Ruder EH, Blumberg J, Hartman TJ, Goldman MB. Antioxidants in reproductive health and fertility. In Al-Gubory KH, Laher I (eds). Nutritional Antioxidant Therapies: Treatments and Perspectives. Springer-Verlag (Germany), in press.
- [Result] Patchell FS, Ruder EH, Mitchell DC, Hartman TJ, Goldman MB. A comparison of energy and antioxidant intake using the Block FFQ and unannounced 24-hour recalls among couples planning pregnancy. 7th International Conference on Diet and Activity Methods, June 4-7, 2009, Washington, DC.
- [Result] Patchell FS, Ruder EH, Mitchell DC, Jacques PF, Hartman TJ, Goldman MB. A comparison of selected nutrient intakes between the Block FFQ and unannounced 24-hour dietary recalls in periconceptional couples. Experimental Biology, Washington, DC, April 9-13, 2011.
- [Result] Ruder EH, Hartman TJ, Reindollar RH, Goldman MB. Female dietary antioxidant intake and time to pregnancy among couples treated for unexplained infertility. Fertil Steril. 2014 Mar;101(3):759-66. doi: 10.1016/j.fertnstert.2013.11.008. Epub 2013 Dec 17. PMID 24355050
- [Result] Pacis MM, Goldman MB, Fung JL, Reindollar RH. Is there an association between Vitamin D intake and time to conception? Data from the FASTT trial. American Society for Reproductive Medicine, Boston, MA, October 12-17, 2013.
- [Result] Hsiao PY, Fung JL, Mitchell DC, Hartman TJ, Goldman MB. Dietary quality in nulliparous women planning pregnancy: results from the ISIS study. Experimental Biology 2015, Boston, MA, March 28-April 1, 2015.
- [Result] Goldman MB, Fung JL, Blumberg J, Hartman TJ. Antioxidant intake, oxidative stress, and pregnancy: results from the lifestyle and fertility study (ISIS). Reprod Sci 2016:23 (Suppl 1);186A.
- [Result] Fung JL, Hartman TJ, Schleicher RL, Goldman MB. Association of vitamin D intake and serum levels with fertility: results from the Lifestyle and Fertility Study. Fertil Steril. 2017 Aug;108(2):302-311. doi: 10.1016/j.fertnstert.2017.05.037. Epub 2017 Jun 16. PMID 28629584
- [Result] Hsiao PY, Fung JL, Mitchell DC, Hartman TJ, Goldman MB. Dietary quality, as measured by the Alternative Healthy Eating Index for Pregnancy (AHEI-P), in couples planning their first pregnancy. Public Health Nutr. 2019 Dec;22(18):3385-3394. doi: 10.1017/S1368980019001290. Epub 2019 May 27. PMID 31131783